CLINICAL TRIAL: NCT03166540
Title: Bioavailability and Beneficial Properties of Espresso Coffee and Confectionery Derived Coffee Bioactive Compounds
Brief Title: Bioavailability and Beneficial Properties of Coffee and Cocoa Bioactive Compounds
Acronym: P4L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Daniele Del Rio, Prof., University of Parma
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DDR-P4L
Record Dates: First submitted 2017-05-21; First posted 2017-05-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Diet Modification; Cardiovascular Risk Factor; Nutritional and Metabolic Diseases
Keywords: coffee; cocoa; bioavailability; pharmacokinetics; cardiometabolic risk factors; caffeoylquinic acids; flavan-3-ol; caffeine; trigonelline; diterpene
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Sample codification, done by the PI, will be hidden to the researchers analysing the samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low consumers (Experimental): 1 cup of espresso coffee/day at 9.00 A.M. for 1 month
  Interventions: Other: cup of espresso coffee
- high consumers (Experimental): 3 cup of espresso coffee/day at 9.00 A.M. 12.00 P.M. and 3.00 P.M. for 1 month
  Interventions: Other: cup of espresso coffee
- medium consumers (Experimental): 1 cup of espresso coffee at 9.00 A.M. + cocoa-based products containing coffee at 12.00 P.M. and 3.00 P.M. for 1 month
  Interventions: Other: cup of espresso coffee; Other: cocoa-based products containing coffee

INTERVENTIONS:
Other: cup of espresso coffee — Subjects will consume the assigned treatment for one month. Espresso coffee will be prepared by using coffee capsules. Serving size: approximately 45 mL. The last day of the intervention is the sampling day.
Other: cocoa-based products containing coffee — Subjects will consume the assigned treatment (2 products per serving) for one month. Serving size: approximately 37 g. The last day of the intervention is the sampling day.
  Arms: medium consumers

SUMMARY:
The aim of this study will be to define the bioavailability and the beneficial properties of coffee bioactive compounds. Moreover, the contribution of cocoa-based products containing coffee to the pool of circulating metabolites will be investigated with the aim of evaluating the effect of the combination of bioactives from different sources.

To study the bioavailability of coffee/cocoa bioactive compounds and their effects in cardiometabolic health, the objectives will be:

i) Assessing the bioavailability of the four main groups of phytochemicals in roasted coffee (methylxanthines, phenolic compounds, trigonelline, and diterpenes), its modulation by the level of consumption, and establishing the daily average concentration of coffee-derived plasma circulating metabolites; ii) Investigating the effect of different levels of coffee consumption on cardiometabolic risk factors; iii) Evaluating circulating metabolites and their putative bioactivity when substituting coffee consumption with the intake of cocoa-based products containing coffee.

A 3-arm, crossover, randomized trial will be conducted. Twenty-one volunteers will be randomly assigned to consume three treatments in a random order for 1 month: 1 cup of espresso coffee/day, 3 cups of espresso coffee/day, 1 cup of espresso coffee at breakfast and 2 cocoa-based products containing coffee two times per day. The last day of the treatment subjects will refer to the ambulatory where blood and urine samples will be collected at specific time points up to 24 hours following the consumption of the testing coffee or of the cocoa-based products containing coffee. In addition to the bioavailability of the bioactive compounds, the effect of the coffee consumption on several cardiometabolic risk factors (blood pressure, anthropometric measures, inflammatory markers, nitric oxide, blood lipids, fasting indices of glucose/insulin metabolism, DNA damage, eicosanoids, nutri-metabolomics) will be investigated. At the end of the treatment, the same protocol will be repeated, switching the allocation group.

DETAILED DESCRIPTION:
A human bioavailability study will be carried out to achieve the above-described goals. The human intervention study will consist of a short-term randomized cross-over trial, addressed at measuring the daily mean concentrations of each coffee/cocoa-derived circulating metabolite (CCDCM) for the four main groups of coffee/cocoa phytochemicals (methylxanthines, trigonelline, phenolics, diterpenes). On the basis of different patterns of consumption, this free-living study (although some minimal dietary restrictions will be provided two days before sampling times) will also take into consideration the effects of repeated doses on the bioavailability of coffee/cocoa bioactives.

The study will follow a repeat-dose, 3-arm, cross-over design. This design has been chosen according to ILSI's guidelines for intervention trials with dietary products.

Subjects were assigned to consume the following treatments in a random order for 1 month:

1. 1 cup of espresso coffee/day ("low consumers") at 9.00 A.M.
2. 3 cups of espresso coffee/day ("high consumers") at 9.00 A.M., 12.00 P.M.noon and 3.00 P.M.
3. 1 cup of espresso coffee at breakfast 9.00 A.M. and 2 cocoa-based products containing coffee two times per day (at 12.00 P.M.noon and 3.00 P.M.). The group will be named "medium consumers", considering the caffeine content of the cocoa-based products containing coffee.

Minimal recommendations to avoid other sources of coffee/cocoa phytochemicals besides what introduced through the assigned treatment, and to standardise the time of coffee consumption, will be provided for the two days prior to each sampling day and on the sampling day. Dinner timing and composition will also be standardised the day before the sampling day. Only water could be drunk during the night. At the sampling day (i.e. the last day of each intervention period), the subjects will refer in the morning at the ambulatory where fasting baseline blood and urine samples will be collected. Then, low and high consumers will drink one or three cups of espresso coffee, respectively (without sugar, sweeteners, and milk for the first coffee; with 5 g of sugar for the last two coffees), while medium consumers will drink a cup of espresso coffee and 2 cocoa-based products containing coffee twice during the day, following the above-described timing. After ingestion of the first coffee together with a phytochemical-free breakfast (a pastry), blood and urine samples will be collected at selected time points along the following 24-h. Five hours after the consumption of the first coffee, participants will receive a standardised mixed meal (sandwich with ham and cheese) free of coffee/cocoa phytochemical-related compounds. Water will be available ad libitum. Twenty-four hours after receiving the treatment, blood and urine samples will also be taken in order to assess return to baseline. In addition, anthropometric characteristics and blood pressure (BP) will be measured.

Socio-demographic variables will be assessed through a generic questionnaire filled at recruitment. The questionnaire will also contain questions useful to identify possible exclusion criteria (e.g. diagnosis for diseases, regular consumption of medication, food allergy). Dietary habits of volunteers will also be evaluated during the enrollment, through a semi-quantitative food frequency questionnaire (FFQ) for the assessment of dietary total antioxidant capacity. In addition, participants' food intakes and compliance with the study requirements will be assessed by means of 3-day dietary records, administered throughout each intervention period at two time points: i) in the middle of each intervention period during two weekdays and a weekend day, and ii) at the end of each intervention period, 2 days prior to the sampling day and the sampling day. The habitual physical activity level of each participant will be measured through a validated International Physical Activity Questionnaires.

Blood sample collection will be carried out in the ambulatory unit of the Department of Medicine and Surgery. Blood collection will be carried out by a physician. A venous catheter will be inserted into the antecubital vein and blood samples from each subject will be collected in specific tubes over 24 hours. Blood sampling at time-point 24h after first coffee consumption will be done by venipuncture. Urine samples will be collected during different periods of time using urine collectors.

Blood samples will be centrifuged and plasma, serum and peripheral blood mononuclear cells (PBMCs) will be collected, aliquoted, and stored at -80 °C for further processing. Urine samples will be aliquoted and stored at -80°C for further processing.

The primary selected endpoint of the study is the quantification of the daily mean concentration of coffee-derived plasma circulating phenolic metabolites, whereas the study of the bioavailability of other coffee-derived circulating bioactives, the bioavailability of cocoa-derived circulating phytochemicals, and the assessment of cardiometabolic markers will be considered secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* adult
* both genders
* healthy
* normal weight (BMI 18-25)
* regular coffee consumers of 1-5 cups per day

Exclusion Criteria:

* younger than 18 y.o. or older than 60 y.o.
* clinically diagnosis for metabolic, renal or digestive disorders
* regular consumption of medication
* antibiotic therapy taken within the last 3 months
* intense physical activity
* pregnancy or lactation
* underweight or overweight/obese
* no regular consumption of coffee or regular intake exceeding 5 coffees/day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Daily mean concentration of phenolic metabolites | 24 hours (0 -overnight fasting-, 30, 60, 120, 180, 240, 300, 360, 420, 480, 540, 1440 -overnight fasting- minutes)
  Assessment of the daily mean concentration of coffee derived plasma circulating phenolic metabolites

SECONDARY OUTCOMES:
Coffee-derived plasma circulating bioactives | 24 hours (0 -overnight fasting-, 30, 60, 120, 180, 240, 300, 360, 420, 480, 540, 1440 -overnight fasting- minutes)
  Profile of metabolites coming from coffee phytochemicals (phenolic compounds, trigonelline, caffeine, and diterpenes) in plasma
Coffee-derived bioactives in urine | 24 hours (0 -overnight fasting-, 180, 360, 540, 1440 -overnight fasting- minutes)
  Profile of metabolites coming from coffee phytochemicals (phenolic compounds, trigonelline, caffeine, and diterpenes) in urine
Cocoa-derived plasma circulating bioactives | 24 hours (0 -overnight fasting-, 30, 60, 120, 180, 240, 300, 360, 420, 480, 540, 1440 -overnight fasting- minutes)
  Profile of metabolites coming from cocoa phytochemicals (phenolic compounds and theobromine) in plasma
Cocoa-derived bioactives in urine | 24 hours (0 -overnight fasting-, 180, 360, 540, 1440 -overnight fasting- minutes)
  Profile of metabolites coming from cocoa phytochemicals (phenolic compounds and theobromine) in urine
Blood Pressure | two time (0 -overnight fasting-, 1 month-fasting-)
  Systolic and diastolic blood pressure
Body Mass Index (BMI) | two time (0 -overnight fasting-, 1 month-fasting-)
  Weight (in kg) and height (in m) will be combined to report BMI in kg/m2
Waist circumference | two time (0 -overnight fasting-, 1 month-fasting-)
Trimethyl-ammine-N-oxide (TMAO) in plasma | 24 hours (0 -overnight fasting-, 30, 60, 120, 180, 240, 300, 360, 420, 480, 540, 1440 -overnight fasting- minutes)
Trimethyl-ammine-N-oxide (TMAO) in urine | 24 hours (0 -overnight fasting-, 180, 360, 540, 1440 -overnight fasting- minutes)
Nitric oxide (NO) in plasma | 1440 -overnight fasting- minutes
Blood lipids | 1440 -overnight fasting- minutes
  Total cholesterol, HDL, LDL, triglycerides
Glucose and Insulin | 1440 -overnight fasting- minutes
  Fasting glucose and fasting insulin
DNA damage | 24 hours (0 -overnight fasting-, 60, 240, 420, 1440 -overnight fasting- minutes)
  Assessed by using the Comet assay
DNA catabolites | 24 hours (0 -overnight fasting-, 60, 240, 420, 1440 -overnight fasting- minutes)
  Assessed by using LC-MS for individual detection and quantification
Nutri-metabolomics in plasma | 1440 -overnight fasting- minutes
  Metabolomics will be carried out in fasting plasma to unravel the potential metabolic pathways of molecules present in the food matrix
Nutri-metabolomics in urine | 24 hours (0 -overnight fasting-, 180, 360, 540, 1440 -overnight fasting- minutes)
  Metabolomics will be carried out in urine to unravel the potential metabolic pathways of molecules present in the food matrix
Eicosanoids in urine | 24 hours (0 -overnight fasting-, 180, 360, 540, 1440 -overnight fasting- minutes)
Inflammatory markers in plasma | 1440 -overnight fasting- minutes
  Main inflammatory markers associated with coffee consumption

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Del Rio, Ph.D., Principal Investigator — University of Parma; Pedro M Mena Parreño, Ph.D., Study Director — University of Parma
Locations (1):
- Department of Food and Drug, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mena P, Bresciani L, Tassotti M, Rosi A, Martini D, Antonini M, Cas AD, Bonadonna R, Brighenti F, Del Rio D. Effect of different patterns of consumption of coffee and a cocoa-based product containing coffee on the nutrikinetics and urinary excretion of phenolic compounds. Am J Clin Nutr. 2021 Dec 1;114(6):2107-2118. doi: 10.1093/ajcn/nqab299. PMID 34582552
- [Derived] Martini D, Rosi A, Tassotti M, Antonini M, Dall'Asta M, Bresciani L, Fantuzzi F, Spigoni V, Dominguez-Perles R, Angelino D, Ricci C, Del Pozo-Luengo S, Tornel PL, Scazzina F, Gil-Izquierdo A, Dei Cas A, Brighenti F, Bonadonna R, Del Rio D, Mena P. Effect of coffee and cocoa-based confectionery containing coffee on markers of cardiometabolic health: results from the pocket-4-life project. Eur J Nutr. 2021 Apr;60(3):1453-1463. doi: 10.1007/s00394-020-02347-5. Epub 2020 Jul 29. PMID 32728879
- [Derived] Mena P, Tassotti M, Martini D, Rosi A, Brighenti F, Del Rio D. The Pocket-4-Life project, bioavailability and beneficial properties of the bioactive compounds of espresso coffee and cocoa-based confectionery containing coffee: study protocol for a randomized cross-over trial. Trials. 2017 Nov 9;18(1):527. doi: 10.1186/s13063-017-2271-2. PMID 29121975